CLINICAL TRIAL: NCT01575288
Title: Oral Trehalose Therapy to Reverse Arterial Aging in Middle-Aged and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B6310
Record Dates: First submitted 2012-04-06; First posted 2012-04-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Vascular Aging
Keywords: arterial function; cardiovascular; aging; endothelial function; arterial stiffness; vascular function; Trehalose
MeSH Terms: interventions — Trehalose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maltose (Placebo Comparator)
  Interventions: Drug: Placebo
- High-dose trehalose (Experimental)
  Interventions: Drug: High-dose trehalose

INTERVENTIONS:
Drug: Placebo — 100g maltose 1/day
  Arms: Maltose
Drug: High-dose trehalose — 100g 1/day
  Arms: High-dose trehalose

SUMMARY:
The proposed study will assess the ability of a naturally occurring sugar to improve the function of arteries with age. Overall, the proposed research project has the long-term potential to influence clinical practice guidelines by establishing a novel, easy to deliver, cost-effective therapy for treating age-associated arterial dysfunction and reducing the risk of cardiovascular disease with age.

ELIGIBILITY:
Inclusion Criteria:

* women must be postmenopausal
* body mass index (BMI) <40 kg/m2
* weight stable in the prior 3 months
* absence of clinical disease as determined by medical history, physical examination, blood and urine chemistries, ankle-brachial index, and a graded exercise stress test with monitoring of blood pressure and 12-lead ECG

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | 12 weeks
  Arterial pulse wave velocity
nitric-oxide mediated endothelium-dependent dilation | 12 weeks
  flow-mediated dilation and forearm blood flow responses to acetylcholine in the presence and absence of N'-monomethyl-L-arginine

SECONDARY OUTCOMES:
Systemic oxidative stress and inflammation | 12 weeks
  circulating markers of oxidative stress and inflammation
Endothelial cell oxidative stress and inflammation | 12 weeks
  inflammatory and oxidative stress markers in biopsied vascular and arterial endothelial cells
Insulin sensitivity | 12 weeks
  intravenous glucose tolerance test
Endothelial cell autophagic flux | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle E Kaplon, MS, Study Director — University of Colorado, Denver; Douglas R Seals, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Boulder Clinical Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- See also: Description of our Research and Laboratory — http://www.colorado.edu/intphys/research/cardiovascular.html